CLINICAL TRIAL: NCT05504434
Title: Performance of a Single-use Gastroscope (aScope Gastro) for Esophagogastroduodenoscopy
Acronym: FARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maag Lever Darm Stichting (Other); Ambu A/S (Industry)
Responsible Party: Principal Investigator, Marco J. Bruno, Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2022-0285
Record Dates: First submitted 2022-07-22; First posted 2022-08-17 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Gastroscopy; Esophagogastroduodenoscopy; Equipment Design; Equipment Contamination / Prevention & Control; Cross Infection / Prevention & Control; Disposable Equipment; Infection Control / Methods
Keywords: Single-use gastroscope; Equipment Contamination; Performance
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Multi-center prospective consecutive observational cases series study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults patients treated with single use gastroscope (Experimental): Patients will be treated with a single-use gastroscope instead of a reusable gastroscope. The procedure will be performed as normal, no additional actions will be performed.
  Interventions: Device: Single-use gastroscope

INTERVENTIONS:
Device: Single-use gastroscope — Adults patients are treated with a single use gastroscope instead of a reusable gastroscope

SUMMARY:
Several infectious outbreaks have been described in the literature as a result of contaminated endoscopes. These endoscopes cannot be sterilized and require an extensive cleaning process in which breaches of cleaning protocols, endoscope damage or the formation of biofilm can prevent proper disinfection. The risk of endoscopy associated infection (EAI) and colonization due to contaminated endoscopes is still considered to be low. However, it is likely that there is severe underreporting of outbreaks due to a lack of recognition or assuming an infection to be endogenous. Due to the sheer volume of upper-gastrointestinal endoscopy worldwide, even with a low risk of EAI, the number of affected patients is significant. In response, several manufacturers have turned to the production of single-use endoscopes that eliminate the risk of exogenous infections. There are single use duodenoscopes on the market that almost seem to match the performance of reusable duodenoscopes. A new single use sterile gastroscope, Ambu aScope gastro, has been developed whose performance has not been previously described in patients. This multicenter single arm consecutive case series study will test the performance of these single use gastroscopes in patients undergoing esophagogastroduodenoscopy.

DETAILED DESCRIPTION:
Esophagogastroduodenoscopy (EGD) is an important tool in the diagnosis and treatment of upper gastrointestinal-disorders. It has broad range of indications including dysphagia, gastroesophageal reflux disease, esophageal strictures or upper gastrointestinal (GI) bleeding. It is a common procedure and is performed around 6.1 million times annually in the United States. However, performing endoscopy is not without risk and complications of EGD include perforation, bleeding, aspiration, and infection.

Endoscopy associated infection (EAI) can be endogenous, due to translocation of the patient's own microbial gut flora into the bloodstream, or exogenous as a result of contaminated equipment. The latter receives increased attention as several outbreaks have been reported past decades. Endoscopes cannot be sterilized and require an extensive cleaning process in which breaches of cleaning protocols, endoscope damage or the formation of biofilm can prevent proper disinfection. Many of the published outbreaks involved contaminated duodenoscopes. However, multiple outbreaks due to a contaminated gastroscopes have also been described. The prevalence of contaminated ready-to-use gastroscopes has rarely been studied. One study reported the contamination of ready-to-use gastroscopes to be 64% post-high-level disinfection (HLD), which went down to 9% post-storage.

It is probable that EAI's are underreported due to a lack of recognition of EAI's caused by sensitive microorganisms, sparse microbiological surveillance post-endoscopy or the possibly long duration between the endoscopy and the development of the infection. However, even if the risk of EAI is low, due to the large numbers of endoscopies performed worldwide the number of affected patients is significant.

Single use endoscopes would completely eliminate the risk of exogenous EAI's. Already multiple single-use duodenoscopes have been brought to the market whose performance seems be comparable to reusable duodenoscopes. To address the risk of contaminated gastroscopes, Ambu is a company who produced a single-use gastroscope, the Ambu® aScope™ gastro. It is a lightweight scope equipped with two LED lights for optimal illumination and a high-resolution digital camera. The aScope gastro has recently been CE-approved, but no studies about its performance in patients have been published

ELIGIBILITY:
Inclusion Criteria:

* Subject is planned to undergo gastroscopy for any indication either outpatient or inpatient
* The subject is ≥ 18 years old

Specifically for the Netherlands:

- The subject is capable to understand the information required to give informed consent

Exclusion Criteria:

* Terminally ill patients
* Patients whose condition in the opinion of the investigator would interfere with adequately assessing the study outcomes
* Patients that participate in other investigational studies which would interfere with the outcomes of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Performance of a single use gastroscope, Ambu aScope gastro, for esophagogastroduodenoscopy | 4 months
  Is the endoscopist able to complete the desired diagnostics/therapeutics during the EGD

SECONDARY OUTCOMES:
Qualitative assessment of the single-use gastroscope | 4 months
  Qualitative assessment of the single-use gastroscope, Ambu aScope gastro, compared to the experience only having used re-usable devices by means of a questionnaire answered by the endoscopist post-EGD. The following characteristics will be rated on a 5 point Likert scale ranging from "much worse" to "much better":
  * Ease of intubation
  * Ease of intubating duodenum
  * Completeness of inspection of the upper digestive track
  * Image quality
  * Handling
  * Lighting
  * Color reproduction
  * Air delivery
  * Therapeutics
Complications of EGD | 4 months
  Complications of EGD including pain post-EGD, bleeding, perforation, and 30-day post-gastroscopy infection rates
Incidence of switching to reusable endoscope | 4 months
Time to complete procedure | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, Professor, Principal Investigator — Erasmus Medical Center
Locations (2):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Oslo University Hospital - Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Ben-Menachem T, Decker GA, Early DS, Evans J, Fanelli RD, Fisher DA, Fisher L, Fukami N, Hwang JH, Ikenberry SO, Jain R, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Dominitz JA, Cash BD. Adverse events of upper GI endoscopy. Gastrointest Endosc. 2012 Oct;76(4):707-18. doi: 10.1016/j.gie.2012.03.252. No abstract available. PMID 22985638
- [Background] McCafferty CE, Aghajani MJ, Abi-Hanna D, Gosbell IB, Jensen SO. An update on gastrointestinal endoscopy-associated infections and their contributing factors. Ann Clin Microbiol Antimicrob. 2018 Oct 10;17(1):36. doi: 10.1186/s12941-018-0289-2. PMID 30314500
- [Background] Ofstead CL, Buro BL, Hopkins KM, Eiland JE, Wetzler HP, Lichtenstein DR. Duodenoscope-associated infection prevention: A call for evidence-based decision making. Endosc Int Open. 2020 Dec;8(12):E1769-E1781. doi: 10.1055/a-1264-7173. Epub 2020 Nov 17. PMID 33269310
- [Background] Bajolet O, Ciocan D, Vallet C, de Champs C, Vernet-Garnier V, Guillard T, Brasme L, Thiefin G, Cadiot G, Bureau-Chalot F. Gastroscopy-associated transmission of extended-spectrum beta-lactamase-producing Pseudomonas aeruginosa. J Hosp Infect. 2013 Apr;83(4):341-3. doi: 10.1016/j.jhin.2012.10.016. Epub 2013 Jan 20. PMID 23337251